CLINICAL TRIAL: NCT05384301
Title: Effects of an Urban Afforestation Activity on Mood, Stress, and Anxiety of Adults
Brief Title: Effects of Urban Afforestation Activity on Mood, Stress, and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, José Manuel Pérez Mármol, Associate Professor, Universidad de Granada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AfforestMood
Record Dates: First submitted 2022-05-17; First posted 2022-05-20 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Healthy
Keywords: Green spaces; Nature-based activities; Urban afforestation; Horticultural therapy; Mental health; Mood; Stress; Anxiety
MeSH Terms: conditions — Psychological Well-Being; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Urban Afforestation Group (Experimental): Participants will perform an afforestation activity with a duration of 90 minutes.
  Interventions: Other: Urban Afforestation Program

INTERVENTIONS:
Other: Urban Afforestation Program — An afforestation program based on land cultivation and transplantation of several plants for 90 minutes will be implemented.
  Other Names: Nature-based activity; Afforestation activity

SUMMARY:
This single-group pretest-posttest clinical trial aims to evaluate the effects of a single-session afforestation activity on mood, stress, and anxiety in a sample of adults.

DETAILED DESCRIPTION:
The participants will perform an afforestation activity for a single session of 90 minutes. The therapist will direct the participants' attention to the visual, auditory, olfactory, and tactile features of the surrounding environment.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18 and 65 years.
* Any sex and gender.

Exclusion Criteria:

* Intake of any psychotropic medication.
* Other severe or medically unstable diseases that may interfere with participation.
* Severe cognitive impairment (Mini-Mental State Examination score < 17 out of 30 points).
* Severe mental disorders in the acute phase or symptomatic phase.
* Severe intellectual disability.
* Behavioural alterations as this may interfere with their participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2022-06-05 (Actual); Study Completion 2022-06-05 (Actual)

PRIMARY OUTCOMES:
Mood | Change from baseline the total mood disturbance after 90 minutes.
  The Spanish adaptation of the 30-item Short Form of the Profile of Mood States will be utilised. There are five questions situated under each mood factor of Anger, Fatigue, Vigour, Friendliness, Tension, and Depressed Mood, which will be rated on a five-point scale starting from 0 indicating "not at all" up to 4 indicating "a lot" to evaluate the current feelings. Higher scores on the vigour and friendliness subscale indicate more positive mood, and higher scores on the remaining subscales indicate more negative mood.

SECONDARY OUTCOMES:
State stress | Change from baseline state stress after 90 minutes.
  The perceived stress will be assessed by the 100-mm Visual Analogue Scale, where endpoints are labelled as "None" and "As bad as it could be" from left to right. The scale will yield a single quantitative variable regarded as the state stress score, which is measured by the distance between the far-left end and the participant's mark on the line in millimetres. Lower scores indicate less stress at the moment.
State anxiety | Change from baseline state anxiety after 90 minutes.
  The 100-mm Visual Analogue Scale for state anxiety will be employed. The endpoints of the scale are labelled as "None" and "As bad as it could be" from left to right. The distance in millimetres between the far-left end and the participant's mark will be regarded as the state anxiety score. Lower scores indicate less anxiety at the moment.

CONTACTS AND LOCATIONS:
Overall Officials: José Manuel PÉREZ-MÁRMOL, PhD, Principal Investigator — Associate Professor
Locations (1):
- University of Granada, Faculty of Health Sciences, Granada, Andalusia, Spain

IPD SHARING:
Plan to Share IPD: No